CLINICAL TRIAL: NCT02997072
Title: Assessment of Regional Lungs Aeration Changes Examined by Impedance Tomography, Depending on the Drive Pressure Applied During High Frequency Jet Ventilation.
Brief Title: Lungs Aeration Changes Examined by Impedance Tomography During High Frequency Jet Ventilation.
Acronym: DPEIT
Status: Completed | Type: Observational
Sponsor: Silesian University of Medicine (Other)
Responsible Party: Principal Investigator, Katarzyna Rybczyk, Principal Investigator, Silesian University of Medicine
Other Study IDs: SilesianMU-PVA1
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Thoracic Diseases
Keywords: electrical impedance tomography; high frequency jet ventilation; drive pressure
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is attempt to establish optimum drive pressure of high frequency jet ventilation during rigid bronchoscopy to ensure good aeration of the lungs examined by electrical impedance tomography.

DETAILED DESCRIPTION:
The study was performed in the Department of Anaesthesiology and Intensive Therapy in Zabrze.

After application of eligibility criteria 30 patients were enrolled in a prospective, observational study. Each patient received an information about the study and the consent form to carry out the measurement procedures was obtained. The data about sex, age, weight, height, comorbidities, BMI were collected.

Patients were given premedication, midazolam (Sopodorm, ICN Polfa Rzeszow, Poland; doses: weight 80kg - 7.5 mg; weight 80-100kg - 15mg) on hour before projected surgery.

Upon arrival to the operating room patient's basic monitoring was provided: ECG (3 leads), heart rate, noninvasive measurement of blood pressure (NIBP), and pulse oximetry. At the same time, a belt with electrodes was put on a patient to monitor impedance tomography, then an automatical record of the basic parameters of regional lung ventilation was turned on.

The medications used for induction of anesthesia: fentanyl (Fentanyl WZF, Polfa Warsaw, Poland) at a dose of 2 g /kg bw i.v., propofol (Diprivan, AstraZeneca, PolskaPlofed Polpharma Poland) at a dose of 2 mg / kg bw, i.v. and to carry out an intubation - cis-atracurium (Nimbex, GlaxoSmithKine, UK) at dose of 0.15 mg /kg bw i.v. During rigid bronchoscopy maintenance of general anesthesia was achieved through the supply of intravenous propofol at a dose of 10 - 6 mg/kg bw/h.The high frequency jet ventilation (HFJV) was performed with proper respirator (Universal Jet Ventilator Monsoon DeLuxe ACUTRONIC Switzerland), using following ventilation parameters: f = 160-200 breaths / min, FiO2 (fraction of inspired oxygen) = 1, the DP (drive pressure) = 1.5-2.5 Atm. Simultaneously, patients were monitored using a PulmoVista 500 Dräger device and aeration of the lungs examined by electrical impedance tomography were observed in a monitor.

During anesthesia, patients received hydration in the form of a 0.9% solution of Ringer's lactate at 4 ml/kg bw/h. In the event of bradycardia atropine (Atropine sulfuricum, Polfa Warsaw, Poland) at dose of 0.5 mg iv was given, in the event of a decrease in mean arterial pressure below 70 mmHg or 25% compared to the output pressure, ephedrine (Ephedrinum Hydrochloricum WZF, Polfa Warsaw, Poland) in fractionated doses of 5 mg iv (Max 25 mg) was given and in the case of the ineffectiveness of the proceedings dopamine infusion (Dopaminum Hydrochloricum WZF 4%, Polfa Warsaw, Poland) in the syringe pump titrated to maintain a mean arterial pressure above 70 mmHg.

Recovery from anesthesia took place at the recovery room after the removal of the anesthetics and muscle relaxants. If necessary, reverse the action of muscle relaxants was announced neostigmine (Polstygminum, Teva Pharmaceuticals Poland, Poland) at a dose of 0.5 - 2.5 mg i.v.

During anesthesia following parameters were monitored: ECG (3 leads), heart rate, noninvasive blood pressure (NIBP) every 3 minutes and arterial oxygen saturation measured by pulse oximetry.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18
* Obtained written consent form to participate in research
* Patients qualified for rigid bronchoscopy procedure

Exclusion Criteria:

* Absence of the written consent to participate in research
* Undergoing urgent treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group of 30 patients hospitalized in 1st Clinical Hospital in Zabrze that were qualified for planned thoracotomy or videothoracoscopy with the preceding rigid bronchoscopy procedure.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Lung aeration corresponding to each layer of the lungs. | 10 minutes
  The numerical values indicating the percentage of total increased resistance corresponding to each layer of the lungs (ROI - region of interests) that were collected in 15-seconds intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Misiołek, MD, PhD, Prof, Study Chair — School of Medicine with the Division of Dentistry in Zabrze. Medical University of Silesia. Department of Anaesthesiology and Critical Care.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bialka S, Copik M, Rybczyk K, Owczarek A, Jedrusik E, Czyzewski D, Filipowski M, Rivas E, Ruetzler K, Szarpak L, Misiolek H. Assessment of changes of regional ventilation distribution in the lung tissue depending on the driving pressure applied during high frequency jet ventilation. BMC Anesthesiol. 2018 Jul 31;18(1):101. doi: 10.1186/s12871-018-0552-2. PMID 30064377